CLINICAL TRIAL: NCT00685659
Title: Effectiveness of Extended Treatments for Drug Dependence
Acronym: ETDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA020623 (NIH); R01DA020623 (NIH)
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-06

CONDITIONS: Cocaine Dependence
Keywords: cocaine dependence; treatment; continuing care; outcomes; incentives; adaptive
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAU only (Active Comparator): Control condition that consists of treatment as usual, which is Intensive Outpatient Treatment (about 3 months long)
  Interventions: Other: Intensive Outpatient Treatment
- TMAC only (Experimental): Adaptive telephone-based counseling
  Interventions: Other: Adaptive telephone-based counseling
- TMAC plus (Experimental): Adaptive telephone-based counseling, plus incentives
  Interventions: Other: Adaptive telephone-based counseling plus incentives

INTERVENTIONS:
Other: Intensive Outpatient Treatment — 9 hours of group counseling per week for 2-3 months
  Arms: TAU only
Other: Adaptive telephone-based counseling — In addition to IOP, patients receive telephone counseling calls, in which risk level is assessed and coping skills intervention delivered to address risk areas. Adaptive stepped care algorithm is included
  Arms: TMAC only
Other: Adaptive telephone-based counseling plus incentives — In addition to IOP, patients receive telephone counseling calls, in which risk level is assessed and coping skills intervention delivered to address risk areas. Adaptive stepped care algorithm and monetary incentives for participation are included
  Arms: TMAC plus

SUMMARY:
This study tests the effectiveness of two 24 month, telephone-based adaptive continuing care interventions for patients with cocaine dependence. The two interventions are predicted to produce better drug use outcomes than standard care. Furthermore, the intervention that also includes monetary incentives for continued participation is hypothesized to produce better retention and drug use outcomes than the intervention without incentives. Economic analyses will determine the cost-effectiveness and benefit-cost of the interventions relative to standard care, and to each other.

DETAILED DESCRIPTION:
There is considerable evidence that treatment for drug use disorders can lead to substantial improvements in substance use and psychosocial problem severity. However, a significant percentage of patients relapse to problematic levels of substance use after primary treatment, and require additional treatment episodes. Patients are therefore frequently referred to continuing care programs to prevent relapse and decrease the probability of additional rehabilitation treatments. However, current models of continuing care may not be adequate for the long-term management of a chronic, relapsing disorder such as substance dependence. One possible approach for improving the management of drug dependence is adaptive treatment regimes, which combine low intensity monitoring and counseling when patients are doing well with stepped care protocols to increase the intensity of treatment when warranted by deteriorations in status and functioning. However, addiction management protocols may require incentives and other features to make long-term participation more appealing.

Cocaine dependent patients who have completed 2 weeks of intensive outpatient treatment (IOP) will be randomly assigned to one of the following interventions: (1) continued participation in IOP without additional intervention (TAU); (2) TAU plus an adaptive protocol that includes monitoring, feedback, and brief counseling via telephone on a tapered schedule out to 24 months, and more intensive face-to-face treatment when warranted (TMAC); or (3) TAU and the adaptive protocol, plus incentives for sustained participation (TMAC-Plus). Patients will be followed up at 3, 6, 9, 12, 18, and 24 months post intake into the study. Follow-up assessments will include measures of drug use, treatment process and potential mediating factors, psychosocial problem severity, utilization of health and social services, and costs.

The two adaptive extended interventions (TMAC and TMAC-Plus) are predicted to produce better drug use outcomes than TAU. TMAC-Plus is hypothesized to produce better retention and drug use outcomes than TMAC. Economic analyses will determine the cost-effectiveness and benefit-cost of TMAC and TMF-Plus relative to TAU, and to each other. Other analyses will test mediation hypotheses, examine potential moderator effects, and test the impact of disease management on HIV risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* qualify for a DSM-IV lifetime diagnosis of cocaine dependence and cocaine use in 6 months prior to treatment;
* initial engagement in IOP, as indicated by attendance at 4 or more sessions in the first two weeks of treatment;
* 18 to 75 years of age;
* willingness to be randomized and participate in research.
* metropolitan area residents;
* able to provide the name, verified telephone number, and address of at least one contact who can provide locator information on the patient during follow-up.

Exclusion Criteria:

* current psychotic disorder or evidence of dementia severe enough to prevent participation in outpatient treatment;
* acute medical problem requiring immediate inpatient treatment;
* current participation in methadone or other forms of DA treatment, other than IOP

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2007-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R McKay, Ph.D., Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Presbyterian Hospital, Philadelphia, Pennsylvania
  - NorthEast Treatment Centers, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McKay JR, Van Horn DH, Lynch KG, Ivey M, Cary MS, Drapkin ML, Coviello DM, Plebani JG. An adaptive approach for identifying cocaine dependent patients who benefit from extended continuing care. J Consult Clin Psychol. 2013 Dec;81(6):1063-73. doi: 10.1037/a0034265. Epub 2013 Sep 16. PMID 24041231
- [Result] McKay JR, Van Horn DH, Lynch KG, Ivey M, Cary MS, Drapkin M, Coviello D. Who benefits from extended continuing care for cocaine dependence? Addict Behav. 2014 Mar;39(3):660-8. doi: 10.1016/j.addbeh.2013.11.019. Epub 2013 Dec 1. PMID 24355401
- [Result] McKay JR, Van Horn D, Rennert L, Drapkin M, Ivey M, Koppenhaver J. Factors in sustained recovery from cocaine dependence. J Subst Abuse Treat. 2013 Aug;45(2):163-72. doi: 10.1016/j.jsat.2013.02.007. Epub 2013 Apr 2. PMID 23561331
- [Result] Van Horn DH, Drapkin M, Ivey M, Thomas T, Domis SW, Abdalla O, Herd D, McKay JR. Voucher incentives increase treatment participation in telephone-based continuing care for cocaine dependence. Drug Alcohol Depend. 2011 Apr 1;114(2-3):225-8. doi: 10.1016/j.drugalcdep.2010.09.007. Epub 2010 Nov 1. PMID 21041041
- [Result] Wimberly AS, Ivey M, Rennert L, McKay JR. Effect of Continuing Care for Cocaine Dependence on HIV Sex-Risk Behaviors. AIDS Behav. 2017 Apr;21(4):1082-1090. doi: 10.1007/s10461-016-1434-6. PMID 27224980
- [Result] McCollister K, Yang X, McKay JR. Cost-effectiveness analysis of a continuing care intervention for cocaine-dependent adults. Drug Alcohol Depend. 2016 Jan 1;158:38-44. doi: 10.1016/j.drugalcdep.2015.10.032. Epub 2015 Nov 12. PMID 26621551

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled 332, but 11 of those were pilot participants assigned to receive the Telephone Monitoring and Counseling plus vouchers. They were not randomly assigned participants and their data was not included in the final analyses.
Groups:
- Treatment as Usual: Control condition that consists of treatment as usual, which is Intensive Outpatient Treatment (about 3 months long)
  Intensive Outpatient Treatment: 9 hours of group counseling per week for 2-3 months
- TMAC: Adaptive telephone-based counseling
  Adaptive telephone-based counseling: In addition to IOP, patients receive telephone counseling calls, in which risk level is assessed and coping skills intervention delivered to address risk areas. Adaptive stepped care algorithm is included
Period: Overall Study
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Started | 108 | 106 | 107
Completed | 77 | 81 | 92
Not Completed | 31 | 25 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment as Usual | TMAC | TMAC Plus | Total
Number analyzed (Participants) | 108 | 106 | 107 | 321
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (8.0) | 43.3 (7.8) | 43.4 (6.48) | 43.2 (7.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 24 | 76
  Male | 82 | 80 | 83 | 245
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 3 | 12
  Not Hispanic or Latino | 105 | 99 | 104 | 308
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 97 | 89 | 98 | 284
  White | 8 | 10 | 6 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 7 | 3 | 13
Region of Enrollment [Number; unit: participants]
  United States | 108 | 106 | 107 | 321

OUTCOME MEASURES:

1. Primary Outcome: Abstinence
Description: Abstinence as reported on Addiction Severity Index, Timeline Follow up, and as tested on the urine drug screen. Measure was created as such: if on ASI the participant reported no use, and on the TLFB the participant reported no use, and on the urine drug screen there was no substances detected, then the participant is considered abstinent. If there is use indicated on any one or all of those items (ASI, TLFB, UDS) then the participant is not abstinent.
Time Frame: 3 month follow up
Population: The N analyzed represents that number of people we reached for three month follow up evaluation.
Measure: Number; unit: participants
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 96 | 97 | 96
participants | 45 | 57 | 45

2. Primary Outcome: Abstinence
Description: as for outcome 1
Time Frame: 6 month follow up
Population: The N analyzed represents that number of participants we reached for 6 month follow up evaluation.
Measure: Number; unit: participants
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 95 | 95 | 95
participants | 43 | 44 | 42

3. Primary Outcome: Abstinence
Description: as for outcome 1
Time Frame: 9 month follow up
Population: The N analyzed represents the number of participants we were able to reach for the 9 month follow up evaluation.
Measure: Number; unit: participants
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 91 | 91 | 91
participants | 43 | 44 | 39

4. Primary Outcome: Abstinence
Description: as for outcome 1
Time Frame: 12 month follow up
Population: The N analyzed represents the number of participants we were able to reach at the 12 month follow up for evaluation.
Measure: Number; unit: participants
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 89 | 90 | 90
participants | 33 | 39 | 42

5. Primary Outcome: Abstinence
Description: as for outcome 1
Time Frame: 18 month follow up
Population: The N analyzed represents the number of participants we were able to reach for the 18 month follow up.
Measure: Number; unit: participants
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 77 | 79 | 83
participants | 30 | 27 | 34

6. Primary Outcome: Abstinence
Description: as for outcome 1
Time Frame: 24 month follow up
Population: The N analyzed represents the number of participants we were able to reach for 24 month follow up.
Measure: Number; unit: participants
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 59 | 64 | 68
participants | 20 | 28 | 24

7. Primary Outcome: Cocaine Urine Toxicology
Description: Positive cocaine test of urine
Time Frame: 3 month follow up
Population: The N analyzed represents the number of participants for whom we had UDS results in month 3.
Measure: Number; unit: proportion of participants positive
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 89 | 76 | 83
proportion of participants positive | 0.31 | 0.22 | 0.20

8. Primary Outcome: Cocaine Urine Toxicology
Description: Positive cocaine test of urine
Time Frame: 6 month follow up
Population: The N analyzed represents the number of participants for whom we had UDS results in month 6.
Measure: Number; unit: proportion of participants positive
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 82 | 76 | 83
proportion of participants positive | 0.26 | 0.24 | 0.28

9. Primary Outcome: Cocaine Urine Toxicology
Description: Positive cocaine test of urine
Time Frame: 9 month follow up
Population: The N analyzed represents the number of participants for whom we had UDS results in month 9.
Measure: Number; unit: proportion of participants positive
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 74 | 69 | 78
proportion of participants positive | 0.30 | 0.25 | 0.29

10. Primary Outcome: Cocaine Urine Toxicology
Description: Positive cocaine test of urine
Time Frame: 12 month follow up
Population: The N analyzed represents the number of participants for whom we had UDS results in month 12.
Measure: Number; unit: proportion of participants positive
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 76 | 73 | 77
proportion of participants positive | 0.37 | 0.27 | 0.27

11. Primary Outcome: Cocaine Urine Toxicology
Description: Positive cocaine test of urine
Time Frame: 18 month follow up
Population: The N analyzed represents the number of participants for whom we had UDS results in month 18.
Measure: Number; unit: proportion of participants positive
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 67 | 72 | 80
proportion of participants positive | 0.33 | 0.29 | 0.24

12. Primary Outcome: Cocaine Urine Toxicology
Description: Positive cocaine test of urine
Time Frame: 24 month follow up
Population: The N analyzed represents the number of participants for whom we had UDS results in month 24.
Measure: Number; unit: proportion of participants positive
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 69 | 80 | 75
proportion of participants positive | 038 | 0.26 | 0.35

13. Primary Outcome: Comparison Across Groups in Societal Costs
Description: Total savings/spending calculated as the monetary value of days of illegal activity, days experiencing medical problems, days experiencing psychiatric problems, and days in jail captured with the ASI. Presented in 2008 dollars.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 108 | 106 | 107
US Dollars | -1545 (23195) | 1564 (10997) | -191 (20514)

14. Primary Outcome: Net Saving/Spending Comparisons Across Groups From Provider Perspective
Description: Savings minus intervention costs. Presented in 2008 dollars.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 108 | 106 | 107
US Dollars | -1545 (23195) | 1222 (11000) | -750 (20477)

15. Primary Outcome: Net Comparisons of Savings and Spendings Across Groups From Societal Perspective
Description: Savings minus intervention costs. Presented in 2008 dollars.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 108 | 106 | 107
US Dollars | -1545 (23195) | 838 (11018) | -1497 (20414)

16. Secondary Outcome: Participation in Protocol
Description: Percent available sessions completed
Time Frame: 24 months
Population: Participants in TAU did not receive telephone counseling so were not included in these analyses. N's for TMAC and TMAC Plus represent participants who completed orientation.
Measure: Mean (Standard Deviation); unit: percentage of sessions
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 0 | 69 | 82
percentage of sessions |  | 38.8 (31.9) | 67.1 (30.7)

17. Secondary Outcome: HIV Sex Risk Score
Description: Risk score from RAB: Risk Assessment Battery. The RAB is a 41 - item self report developed to study the transmission of HIV. The Risk Assessment Battery generates a drug-risk score and a sex-risk score. For this study, the sex-risk score was used as the outcome measure of sexual behavior that is associated with HIV transmission. The sex-risk score ranges from 0 to 18, with 0 denoting no sex-risk and 18 denoting highest sex-risk. Previous research among drug using populations have found a sex-risk score mean of 6.2.
Time Frame: 12 months
Population: N's represent the participants at 12 months for whom we have a completed RAB (Risk Assessment Battery).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 79 | 74 | 77
units on a scale | 2.9 (2.65) | 2.8 (2.10) | 2.7 (2.23)

18. Secondary Outcome: HIV Sex Risk Score
Description: as for outcome 17
Time Frame: 24 months
Population: N's represent the participants at 24 months for whom we have a completed RAB (Risk Assessment Battery).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 70 | 78 | 77
units on a scale | 2.7 (2.45) | 3 (2.74) | 2.7 (2.56)

19. Primary Outcome: Percent Days Cocaine Use
Description: Percent of days during the follow up that there was any cocaine use
Time Frame: 3 months (approximately study days 1 - 90)
Population: N's represent the participants at three months for whom complete Time Line Follow Back data was available.
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 99 | 97 | 97
percentage of days | 4.50 (1.53) | 4.25 (1.56) | 5.91 (1.80)

20. Primary Outcome: Percent Days Cocaine Use
Description: Percent of days during the follow up that there was any cocaine use
Time Frame: 6 months (approproximately study days 91 - 180)
Population: N's represent the participants at three months for whom complete Time Line Follow Back data was available.
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 98 | 91 | 94
percentage of days | 6.60 (1.98) | 7.01 (2.14) | 11.66 (2.47)

21. Primary Outcome: Percent Days Cocaine Use
Description: Percent of days during the follow up that there was any cocaine use
Time Frame: 9 months (approximately study days 181 - 270)
Population: N's represent the participants at three months for whom complete Time Line Follow Back data was available.
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 93 | 87 | 91
percentage of days | 6.96 (2.19) | 8.23 (2.22) | 5.43 (1.81)

22. Primary Outcome: Percent Days Cocaine Use
Description: Percent of days during the follow up that there was any cocaine use
Time Frame: 12 months (approximately study days 271 - 365)
Population: N's represent the participants at three months for whom complete Time Line Follow Back data was available.
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 91 | 87 | 91
percentage of days | 5.58 (1.82) | 8.88 (2.38) | 7.89 (2.37)

23. Primary Outcome: Percent Days Cocaine Use
Description: Percent of days during the follow up that there was any cocaine use
Time Frame: 18 months (approximately study days 366 - 546)
Population: N's represent the participants at three months for whom complete Time Line Follow Back data was available.
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 81 | 82 | 84
percentage of days | 5.13 (1.66) | 6.97 (1.98) | 5.18 (1.48)

24. Primary Outcome: Percent Days Cocaine Use
Description: Percent of days during the follow up that there was any cocaine use
Time Frame: 24 months (approximately study days 547 - 730)
Population: N's represent the participants at three months for whom complete Time Line Follow Back data was available.
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 77 | 82 | 80
percentage of days | 9.80 (2.69) | 6.14 (2.06) | 6.01 (1.77)

25. Primary Outcome: Percent Days Abstinent
Description: Percent of days during the follow up that participant was abstinent from Alcohol and Cocaine
Time Frame: 3 months (approximately study days 1 - 90)
Population: N's represent the participants at three months for whom complete Time Line Follow Back data was available.
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 99 | 97 | 97
percentage of days | 94.01 (1.66) | 89.85 (2.45) | 92.70 (1.85)

26. Primary Outcome: Percent Days Abstinent
Description: Percent of days during the follow up that participant was abstinent from Alcohol and Cocaine
Time Frame: 6 months (approximately study days 91 - 180)
Population: N's represent the participants at three months for whom complete Time Line Follow Back data was available.
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 98 | 91 | 94
percentage of days | 90.20 (2.23) | 89.44 (2.41) | 85.61 (2.75)

27. Primary Outcome: Percent Days Abstinent
Description: Percent of days during the follow up that participant was abstinent from Alcohol and Cocaine
Time Frame: 9 months (approximately study days 181 - 270)
Population: N's represent the participants at three months for whom complete Time Line Follow Back data was available.
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 93 | 87 | 91
percentage of days | 88.16 (2.75) | 87.94 (2.64) | 91.79 (2.08)

28. Primary Outcome: Percent Days Abstinent
Description: Percent of days during the follow up that participant was abstinent from Alcohol and Cocaine
Time Frame: 12 months (approximately study days 271 - 365)
Population: N's represent the participants at three months for whom complete Time Line Follow Back data was available.
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 91 | 87 | 91
percentage of days | 88.91 (2.55) | 87.53 (2.68) | 89.60 (2.50)

29. Primary Outcome: Percent Days Abstinent
Description: Percent of days during the follow up that participant was abstinent from Alcohol and Cocaine
Time Frame: 18 months (approximately days 366 - 546)
Population: N's represent the participants at three months for whom complete Time Line Follow Back data was available.
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 81 | 82 | 84
percentage of days | 86.40 (3.03) | 88.58 (2.55) | 90.56 (1.96)

30. Primary Outcome: Percent Days Abstinent
Description: Percent of days during the follow up that participant was abstinent from Alcohol and Cocaine
Time Frame: 24 months (approximately study days 547 - 730)
Population: N's represent the participants at three months for whom complete Time Line Follow Back data was available.
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
Number analyzed (Participants) | 77 | 82 | 80
percentage of days | 84.00 (3.45) | 88.88 (2.69) | 89.66 (2.42)

ADVERSE EVENTS:
Arm/Group | Treatment as Usual | TMAC | TMAC Plus
All-Cause Mortality (participants affected / at risk) | 2/108 | 1/106 | 1/107
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/106 | 0/107
Other Adverse Events (participants affected / at risk) | 0/108 | 0/106 | 0/107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No